CLINICAL TRIAL: NCT02657122
Title: A Double-blinded, Randomized, Placebo-controlled, Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TD-1473 in Healthy Subjects
Brief Title: SAD and MAD Study to Evaluate Safety, Tolerability, and Pharmacokinetics (PK) of TD-1473 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 0140
Record Dates: First submitted 2015-11-25; First posted 2016-01-15 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Single ascending dose; SAD; multiple ascending dose; MAD; Phase 1; first-in-human; volunteers; TD-1473
MeSH Terms: interventions — izencitinib; Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- TD-1473 for SAD (Experimental): 6 of out 8 subjects per cohort will be randomized to receive TD-1473
  Interventions: Drug: TD-1473 for SAD
- Placebo for SAD (Placebo Comparator): 2 of out 8 subjects per cohort will be randomized to receive placebo
  Interventions: Drug: Placebo for SAD
- TD-1473 for MAD (Experimental): 6 of out 8 subjects per cohort will be randomized to receive TD-1473
  Interventions: Drug: TD-1473 for MAD
- Placebo for MAD (Placebo Comparator): 2 of out 8 subjects per cohort will be randomized to receive placebo
  Interventions: Drug: Placebo for MAD

INTERVENTIONS:
Drug: TD-1473 for SAD — SAD: Healthy subjects meeting eligibility criteria will be sequentially randomized to each dose cohort (up to 5 dose ascending cohorts) to receive either TD-1473 or placebo. The study drug (TD-1473 or placebo) will be administered orally as a single dose.
  Arms: TD-1473 for SAD
Drug: Placebo for SAD — SAD: Healthy subjects meeting eligibility criteria will be sequentially randomized to each dose cohort (up to 5 dose ascending cohorts) to receive either TD-1473 or placebo. The study drug (TD-1473 or placebo) will be administered orally as a single dose.
  Arms: Placebo for SAD
Drug: TD-1473 for MAD — MAD: Healthy subjects meeting eligibility criteria will be sequentially randomized to each dose cohort (up to 4 cohorts) to receive either TD-1473 or placebo. The study drug (TD-1473 or placebo) will be administered orally for a total of 14 days of dosing.
  Arms: TD-1473 for MAD
Drug: Placebo for MAD — MAD: Healthy subjects meeting eligibility criteria will be sequentially randomized to each dose cohort (up to 4 cohorts) to receive either TD-1473 or placebo. The study drug (TD-1473 or placebo) will be administered orally for a total of 14 days of dosing.
  Arms: Placebo for MAD

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of single ascending doses and multiple ascending doses of the investigational drug TD-1473 compared to placebo in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female 19 to 55 years old
* Willing and able to give informed consent
* Body Mass Index (BMI) 18 to 30 kg/m2
* Women of child bearing potential must have a negative pregnancy test and either abstain from sex or use a highly effective method of birth control
* Additional inclusion criteria apply

Exclusion Criteria:

* Positive for hepatitis A, B, or C, HIV, or tuberculosis (TB)
* Clinically significant abnormalities in baseline results of laboratory evaluations
* Evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease
* Participated in another clinical trial of an investigational drug (or medical device) within 30 days prior to Screening (or within 60 days prior to Screening if investigational drug was a biologic), or is currently participating in another trial of an investigational drug (or medical device)
* Use of prescription drugs or any chronic over the counter medications within 14 days prior to clinic admission or requires continuing use during study participation, with the exception of hormonal contraceptives or hormone replacement therapy.
* Additional exclusion criteria apply

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of SAD and MAD of TD-1473 in healthy subjects by assessing the number, severity and type of adverse events, including changes in vital signs, physical examinations, laboratory safety tests and ECGs | Day 1 through Day 8 (SAD) or 21 (MAD)

SECONDARY OUTCOMES:
Area under curve (AUC) in plasma, urine and feces | Day 1 through Day 4-6 (SAD)
Cmax in plasma, urine and feces | Day 1 through Day 4-6 (SAD)
Tmax in plasma, urine and feces | Day 1 through Day 4-6 (SAD)
Terminal elimination half-life (t1/2) in plasma, urine and feces | Day 1 through Day 4-6 (SAD)
Amount excreted in urine (Aeu) | Day 1 through Day 4-6 (SAD)
Amount excreted in feces (Aef) | Day 1 through Day 4-6 (SAD)
AUC in plasma, urine and feces | Day 1 through Day 17-19 (MAD)
Cmax in plasma, urine and feces | Day 1 through Day 17-19 (MAD)
Tmax in plasma, urine and feces | Day 1 through Day 17-19 (MAD)
t1/2 in plasma, urine and feces | Day 1 through Day 17-19 (MAD)
Aeu | Day 1 through Day 17-19 (MAD)
Aef | Day 1 through Day 17-19 (MAD)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

REFERENCES:
- [Derived] Sandborn WJ, Nguyen DD, Beattie DT, Brassil P, Krey W, Woo J, Situ E, Sana R, Sandvik E, Pulido-Rios MT, Bhandari R, Leighton JA, Ganeshappa R, Boyle DL, Abhyankar B, Kleinschek MA, Graham RA, Panes J. Development of Gut-Selective Pan-Janus Kinase Inhibitor TD-1473 for Ulcerative Colitis: A Translational Medicine Programme. J Crohns Colitis. 2020 Sep 16;14(9):1202-1213. doi: 10.1093/ecco-jcc/jjaa049. PMID 32161949